CLINICAL TRIAL: NCT04099953
Title: Atılım University, Physiotherapy and Rehabilitation Department
Brief Title: Does Hemodialysis Affect Upper Extremity Functional Capacity, Physical Activity and Physical Function of Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NAİME ULUG (Other)
Responsible Party: Sponsor-Investigator, NAİME ULUG, Physiotherapist, PhD, Associate Professor, Atılım University
Organization: Atılım University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23/23
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Chronic Kidney Diseases
Keywords: Hemodialysis; chronic renal failure; upper extremity; physical activity; physical function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Motor Activity | interventions — Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dialysis patients (Experimental): Dialysis patients were evaluated by objective diagnostic tests.
  Interventions: Diagnostic Test: Hand grip, joint range of motion , functional level of the upper extremity, physical activity levels
- Control group (Experimental): Healthy individuals
  Interventions: Diagnostic Test: Hand grip, joint range of motion , functional level of the upper extremity, physical activity levels

INTERVENTIONS:
Diagnostic Test: Hand grip, joint range of motion , functional level of the upper extremity, physical activity levels — Hand grip force with Jamar Hand Dynamometer, joint range of motion with Baseline Digital Goniometer, functional level of the upper extremity with the Shoulder-Arm and Hand Problems Questionnaire(DASH), physical activity levels with International Physical Activity Questionnaire Short Form(IPAQ-short form) and physical functions with Human Activity Profile (HAP) were evaluated.

SUMMARY:
This study was planned to determine the effects of upper extremity functional capacity, physical activity level and physical functions of patients receiving hemodialysis treatment.

DETAILED DESCRIPTION:
Upper extremity functional capacity, physical activity level and physical functions were evaluated in healthy subjects and hemodialysis patients.

ELIGIBILITY:
Inclusion criteria:

In study group,

* with cooperation
* hemodialysis treatment for at least 3 months
* with single-sided fistula

In the control group,

* healthy volunteers with no history of trauma or surgery in the upper extremity,
* with cooperating

Exclusion Criteria:

* Individuals with orthopedic problems associated with chronic renal failure,
* Upper limb functions affected

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of The Upper Extremity Functional Level | Evaluations were made after hemodialysis patients rested for half an hour after treatment.
  Turkish version of the Shoulder, Arm and Hand Problems Questionnaire (The DASH-T) was used to asses the functional level of the upper extremity. Turkish version of the shoulder, arm and hand problems questionnaire consists of 30 questions. The first 20 questions are to examine physical competence, and the last 10 questions question pain and related functional and environmental constraints. As the score is closer to zero, the functional level of the person is high; as the score is far from zero the functional level of the person is low .

SECONDARY OUTCOMES:
Evaluation of Physical Activity Level | Evaluations were made after hemodialysis patients rested for half an hour after treatment.
  To asses the level of physical activity, The Turkish version of International Physical Activity Questionnaire Short Form was used . In the turkish version of international physical activity questionnaire short form, physical activities were made at least 10 minutes at a time. In the last 7 days of the survey; Severe physical activity duration (min), moderate physical activity duration (min), walking and one day sitting time (min) were questioned. According to the total physical activity score, the physical activity levels of the participants were classified as low level (under 600 MET min /week), intermediate level (600-3000 MET-min /week) and high level (over 3000 MET-min / week) .
Evaluation of Physical Function Level | Evaluations were made after hemodialysis patients rested for half an hour after treatment.
  The Human Activity Profile (HAP) was used to measure the physical function level. Human activity profile is a scale consisting of 94 items developed to determine the level of physical function in healthy individuals or individuals with chronic diseases at different ages . For each of the 94 items the respondent is asked to indicate whether they are still doing the activity, stopped doing the activity or have never done the activity before. Two scores are calculated: the maximum activity score (MAS) and the adjusted activity score (AAS).
  The physical activity level of the person is in one of 3 subgroups according to the adjusted activity score: <53 points: insufficient activity level, 53-74 points: moderately active and > 74 points: active .

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Cansu AKTAŞ, MsC, Principal Investigator — Atılım University
Locations (1):
- Atılım University, Gölbaşı, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No